CLINICAL TRIAL: NCT06087562
Title: Interspace Between the Popliteal Artery and Capsule of the Posterior Knee (iPACK) Block for Postoperative Rehabilitation in Total Knee Arthroplasty: a Randomized Control Trial
Brief Title: iPACK Block for Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 495/20
Record Dates: First submitted 2023-02-19; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Disease
Keywords: iPACK block; regional anesthesia; multimodal analgesia; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be randomized to one of two groups with a computer-generated arm assignment. The sealed envelopes will be opened immediately before the nerve block. One group will receive an iPACK block, and the other will receive a placebo block. The provider performing the league will not be blinded. However, all other care team members, the patient, and the investigator collecting data will be blinded to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preop iPACK block (Experimental): Patients will receive a preoperative ultrasound-guided Interspace between the Popliteal Artery and Capsule of the Posterior Knee (iPACK) block with 20 mL 0.5% ropivacaine. Using appropriate sterile precautions, and procedural sedation with up to 2 mg IV midazolam, an ultrasound (Mindray TE9) equipped with either a linear 15-6 megahertz (MHz), or a curvilinear 5-2 MHz transducer (habitus-dependent) used to identify the distal femoral shaft and popliteal artery. After spinal anesthesia, a 22g 80 mm echogenic block needle (Stimuplex Ultra 360) is advanced lateral to medial, in-plane, from the anteromedial aspect of the knee, toward the space between the popliteal artery and femur. 20 mL 0.5% ropivacaine is injected into the space between the popliteal artery and femur. The needle is withdrawn, and the needle entry site is wiped clean.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution 20mL
- preop placebo block (Experimental): Patients will receive a preoperative ultrasound-guided Interspace between the Popliteal Artery and Capsule of the Posterior Knee (iPACK) block with 20 mL 0.5% ropivacaine. Using appropriate sterile precautions, and procedural sedation with up to 2 mg IV midazolam, an ultrasound (Mindray TE9) equipped with either a linear 15-6 megahertz (MHz), or a curvilinear 5-2 MHz transducer (habitus-dependent) used to identify the distal femoral shaft and popliteal artery. After spinal anesthesia, a 22g 80 mm echogenic block needle (Stimuplex Ultra 360) is advanced lateral to medial, in-plane, from the anteromedial aspect of the knee, toward the space between the popliteal artery and femur. 20 mL 0.9% normal saline is injected into the space between the popliteal artery and femur. The needle is withdrawn, and the needle entry site is wiped clean.
  Interventions: Drug: 0,9% normal saline 20mL

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution 20mL — Ultrasound-guided iPACK block with 20mL of 0,5% ropivacaine
  Other Names: Ropimol
  Arms: preop iPACK block
Drug: 0,9% normal saline 20mL — Ultrasound-guided placebo block with 20mL of 0,9% normal saline
  Other Names: placebo
  Arms: preop placebo block

SUMMARY:
This randomized, double-blinded, placebo-controlled trial seeks to evaluate the efficacy of the rehabilitation process of the Interspace between the Popliteal Artery and Capsule of the Posterior Knee (iPACK) block in total knee arthroplasty.

DETAILED DESCRIPTION:
The Interspace between the Popliteal Artery and Capsule of the Posterior Knee (iPACK) block, has been recently described and shows promise in providing analgesia to the knee joint. The effect of this block on postoperative rehabilitation is uncertain. This study aims to compare a preoperative iPACK block to a placebo block prior to total knee arthroplasty under spinal anesthesia. The primary outcome measure is verticalization, walking distance, ability to go out of bed, active lifting of the limb, range of motion in the hip joint, bending range of motion, and abduction range of motion. The secondary measure is postoperative pain assessment during rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old undergoing unilateral total knee arthroplasty

Exclusion Criteria:

* refusal to participate
* < 18 yo
* Chronic opioid use
* localized infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale [Range from 0:no pain to 10:the worst pain] | within 24 hours postoperatively
  Numerical Rating Scale [Range from 0:no pain to 10:the worst pain]
Numerical Rating Scale [Range from 0:no pain to 10:the worst pain] | 1 st postoperative day
  NRS (numerical rating scale from 0- no pain to 10- the worst pain)
Numerical Rating Scale [Range from 0:no pain to 10:the worst pain] | 2nd postoperative day
  NRS (numerical rating scale from 0- no pain to 10- the worst pain)
Numerical Rating Scale [Range from 0:no pain to 10:the worst pain] | 5 th postoperative day
  NRS (numerical rating scale from 0- no pain to 10- the worst pain)
Opioid consumption 24 hours postoperatively | 24 hours postoperatively
  intravenous morphine equivalents (mg)
Opioid consumption 48 hours postoperatively | 24-48 hours postoperatively
  intravenous morphine equivalents (mg)
Opioid consumption 72 hours postoperatively | 48-72 hours postoperatively
  intravenous morphine equivalents (mg)
Opioid consumption >72 hours postoperatively | 72-96 hours postoperatively
  intravenous morphine equivalents (mg)
Time to first opioid administration | 0-12 hours postoperatively
  hours

SECONDARY OUTCOMES:
Rehabilitation process Verticalization by the balcony | 1st postoperative day
  Verticalization by the balcony (binary outcome yes or no)
Rehabilitation process Verticalization by the balcony | 2nd postoperative day
  Verticalization by the balcony (binary outcome yes or no)
Rehabilitation process Verticalization by the balcony | 5th postoperative day
  Verticalization by the balcony (binary outcome yes or no)
Rehabilitation process Verticalization with help | 1st postoperative day
  Verticalization- with help (yes/no)
Rehabilitation process Verticalization with help | 2nd postoperative day
  Verticalization- with help (yes/no)
Rehabilitation process Verticalization with help 5th day | 5th postoperative day
  Verticalization- with help (yes/no)
Rehabilitation process Verticalization - impossible 1st day | 1st postoperative day
  Verticalization- impossible (yes/no)
Rehabilitation process Verticalization - impossible 2nd day | 2nd postoperative day
  Verticalization- impossible (yes/no)
Rehabilitation process Verticalization - impossible 5th day | 5th postoperative day
  Verticalization- impossible (yes/no)
Rehabilitation process Walking distance- unlimited with crutches 1st day | 1st postoperative day
  Walking distance- unlimited with crutches (yes/no)
Rehabilitation process Walking distance- unlimited with crutches 2nd day | 2nd postoperative day
  Walking distance- unlimited with crutches (yes/no)
Rehabilitation process Walking distance- unlimited with crutches 5th day | 5th postoperative day
  Walking distance- unlimited with crutches (yes/no)
Rehabilitation process Walking distance- by the balcony 1st day | 1st postoperative day
  Walking distance- by the balcony (yes/no)
Rehabilitation process Walking distance- by the balcony 2nd day | 2nd postoperative day
  Walking distance- by the balcony (yes/no)
Rehabilitation process Walking distance- by the balcony 5th day | 5th postoperative day
  Walking distance- by the balcony (yes/no)
Rehabilitation process Walking distance- impossible- bed bound 1st day | 1st postoperative day
  Walking distance- impossible- bed bound (yes/no)
Rehabilitation process Walking distance- impossible- bed bound 2nd day | 2nd postoperative day
  Walking distance- impossible- bed bound (yes/no)
Rehabilitation process - getting out of bed- no problems 1st day | 1st postoperative day
  getting out of bed with no problems (yes/no)
Rehabilitation process - getting out of bed- no problems 2nd day | 2nd postoperative day
  getting out of bed with no problems (yes/no)
Rehabilitation process - getting out of bed- no problems 5th day | 5th postoperative day
  getting out of bed with no problems (yes/no)
Rehabilitation process - getting out of bed- with help 1st day | 1st postoperative day
  getting out of bed with help (yes/no)
Rehabilitation process - getting out of bed- with help 2nd day | 2nd postoperative day
  getting out of bed with help (yes/no)
Rehabilitation process - getting out of bed- with help 5th day | 5th postoperative day
  getting out of bed with help (yes/no)
Rehabilitation process - getting out of bed- with assistance 1st day | 1st postoperative day
  getting out of bed with assistance (yes/no)
Rehabilitation process - getting out of bed- with assistance 2nd day | 2nd postoperative day
  getting out of bed with assistance (yes/no)
Rehabilitation process - getting out of bed- with assistance 5th day | 5th postoperative day
  getting out of bed with assistance (yes/no)
Rehabilitation process - RANGE OF MOTION - CONTRACTURE IN THE KNEE JOINT - full extension- 1st day | 1st day postoperative day
  CONTRACTURE IN THE KNEE JOINT - full extension (yes/no)
Rehabilitation process - RANGE OF MOTION - CONTRACTURE IN THE KNEE JOINT - full extension- 2nd day | 2nd day postoperative day
  CONTRACTURE IN THE KNEE JOINT - full extension (yes/no)
Rehabilitation process - RANGE OF MOTION - CONTRACTURE IN THE KNEE JOINT - full extension- 5th day | 5th day postoperative day
  CONTRACTURE IN THE KNEE JOINT - full extension (yes/no)
Rehabilitation process - RANGE OF MOTION - flexion contracture IN THE KNEE JOINT - full extension- 1st day | 1st day postoperative day
  flexion contracture IN THE KNEE JOINT (yes/no)
Rehabilitation process - RANGE OF MOTION - flexion contracture IN THE KNEE JOINT - full extension- 2nd day | 2nd day postoperative day
  flexion contracture IN THE KNEE JOINT (yes/no)
Rehabilitation process - RANGE OF MOTION - flexion contracture IN THE KNEE JOINT - full extension- 5th day | 5th day postoperative day
  flexion contracture IN THE KNEE JOINT (yes/no)
Rehabilitation process - bending range of motion- passive movement to 45 degrees- no pain- 1st day | 1st day postoperative day
  bending range of motion- passive movement to 45 degrees with no pain- (yes/no)
Rehabilitation process - bending range of motion- passive movement to 45 degrees- with pain- 1st day | 1st day postoperative day
  bending range of motion- passive movement to 45 degrees with pain- (yes/no)
Rehabilitation process - bending range of motion- passive movement to 45 degrees- no pain- 2nd day | 2nd day postoperative day
  bending range of motion- passive movement to 45 degrees with no pain- (yes/no)
Rehabilitation process - bending range of motion- passive movement to 45 degrees- with pain- 2nd day | 2nd day postoperative day
  bending range of motion- passive movement to 45 degrees with pain- (yes/no)
Rehabilitation process - bending range of motion- passive movement to 45 degrees- no pain- 5th day | 5th day postoperative day
  bending range of motion- passive movement to 45 degrees with no pain- (yes/no)
Rehabilitation process - bending range of motion- passive movement to 45 degrees- with pain- 5th day | 5th day postoperative day
  bending range of motion- passive movement to 45 degrees with pain- (yes/no)
Rehabilitation process - bending range of motion- active movement to 90 degrees- no pain- 5th day | 1st day postoperative day
  bending range of motion- active movement to 90 degrees with no pain- (yes/no)
Rehabilitation process - bending range of motion- active movement to 90 degrees- no pain- 2nd day | 2nd day postoperative day
  bending range of motion- active movement to 90 degrees with no pain- (yes/no)
Rehabilitation process - bending range of motion- active movement to 90 degrees- no pain- 1st day | 1st day postoperative day
  bending range of motion- active movement to 90 degrees with no pain- (yes/no)
Rehabilitation process - bending range of motion- active movement to 90 degrees- with pain- 1st day | 1st day postoperative day
  bending range of motion- active movement to 90 degrees with pain- (yes/no)
Rehabilitation process - bending range of motion- active movement to 90 degrees- with pain- 2nd day | 2nd day postoperative day
  bending range of motion- active movement to 90 degrees with pain- (yes/no)
Rehabilitation process - bending range of motion- active movement to 90 degrees- with pain- 5th day | 5th day postoperative day
  bending range of motion- active movement to 90 degrees with pain- (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Domagalska, PhD, Principal Investigator — Department of Palliative Medicine, University of Medical Sciences, Poznań, Poland; Zbigniew Żaba, PhD, Study Chair — Department of Emergency Medicine
Locations (1):
- Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2024
Access Criteria: The data presented in this study are available on request from the corresponding author.